CLINICAL TRIAL: NCT03347253
Title: A Prospective Study in Subjects With Late Onset Pompe Disease Who Are Currently Being Treated With Enzyme Replacement Therapy
Brief Title: STRIDE Study - A Study in Subjects With LOPD Who Are Currently Being Treated With ERT
Status: Terminated | Type: Observational
Why Stopped: As a result of change of clinical development plan.
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: POM-003
Record Dates: First submitted 2017-11-09; First posted 2017-11-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Late-onset Pompe Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the study is to evaluate changes in key clinical outcome measures (eg, motor, respiratory, fatigue) in adult subjects with late-onset Pompe disease (LOPD) subjects receiving standard-of-care enzyme replacement therapy (ERT). Additionally, information gained may be used in the design and conduct of future studies in LOPD subjects.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the baseline characteristics and degree of change over time in clinical outcome measures commonly used to evaluate patients with LOPD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a diagnosis of Pompe disease based on documented deficiency of GAA activity and a documented GAA mutation.
2. Male and female subjects between 18 years and 75 years, inclusive and ≥ 50 kg.
3. Subject must be currently receiving standard-of-care ERT (alglucosidase alfa) at a dose of 20 mg/kg dose every other week.
4. Subject must have been on ERT for the preceding 2 years or more.
5. Subject must have an upright forced vital capacity (FVC) within 35 to 90% of predicted normal (NHANES III reference values), based on the higher of the screening or baseline value, if their 6 minute walk distance (6MWD) is > 200 m. Subject must have an upright FVC within 40 to 90% of predicted normal (NHANES III reference values), based on the higher of the screening or baseline value, if their 6MWD is ≤ 200 m. If FVC is between 80 and 90% of predicted normal, the subject may enter the study if the percent predicted FVC value drops by 10% predicted or more in supine position
6. Subject is able to walk at least 100 m in the 6MWT and the assessment is noted as valid.

Exclusion Criteria:

1. Subject has received any investigational therapy or pharmacological treatment for Pompe disease, other than alglucosidase alfa within 30 days or 5 half lives, whichever is shorter, prior to the Baseline Visit or is anticipated to do so during the course of the study
2. Subject is on any of the following prohibited medications within 30 days of baseline:

   * miglitol (eg, Glyset)
   * miglustat (eg, Zavesca)
   * acarbose (eg, Precose, Glucobay)
   * voglibose (eg, Volix, Vocarb, Volibo)
3. Subject requires use of invasive or non-invasive ventilatory support for > 6 hours a day while awake.
4. Subject has a medical or any other extenuating condition or circumstance that may, in the opinion of the investigator, pose an undue safety risk to the subject or compromise his/her ability to comply with protocol requirements. This includes clinical depression (as diagnosed by a psychiatrist or other mental health professional) with uncontrolled or poorly controlled symptoms.
5. Subject is breastfeeding, or is pregnant or planning to become pregnant within the next 2 years.
6. Other exclusion criteria according to the Lumizyme/Myozyme instructions for use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects with LOPD between 18 years and 75 years, inclusive and ≥ 50 kg.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate degree of change in muscle function and respiratory endpoints over time | 6-15 month
  To evaluate the degree of change in muscle function and respiratory endpoints over time in patients with Late Onset Pompe disease

CONTACTS AND LOCATIONS:
Locations (21):
- United States (17):
  - University of California, Irvine, Irvine, California
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Emory University, Decatur, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jacobs & Levy Genomic Medicine and Research Program, Morristown, New Jersey
  - Northwell Health, Great Neck, New York
  - NYU Neurogenetics, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health& Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center San Antonio, San Antonio, Texas
- Royal Adelaide Hospital, Adelaide, Australia
- Antwerp University Hospital, Edegem, Belgium
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - McMaster University Medical Center, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No